CLINICAL TRIAL: NCT07206797
Title: Ultrasound for Quantifying Muscle Activation Elicited by Spinal Cord Stimulation and Functional Electrical Stimulation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: North Carolina State University (Other)
Collaborators: University of North Carolina, Chapel Hill (Other)
Responsible Party: Principal Investigator, Nitin Sharma, Principal Investigator, North Carolina State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 24815
Record Dates: First submitted 2025-09-26; First posted 2025-10-03 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Neuromodulatory Effects of TSCS and FES in Lower Limbs
Keywords: Ultrasound; Spinal Stimulation; Functional Electrical Stimulation
MeSH Terms: interventions — Spinal Cord Stimulation; Ultrasonography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Subjects without Disability (Experimental): Up to 30 participants with no disabilities will be recruited.
  Interventions: Device: Functional Electrical Stimulation; Device: Transcutaneous (Non-Invasive) Spinal Cord Stimulation; Device: Ultrasound

INTERVENTIONS:
Device: Functional Electrical Stimulation — Functional electrical stimulation will be applied to the ankle muscles. The resulting torque will be collected, and ultrasound data will be obtained during stimulation.
Device: Transcutaneous (Non-Invasive) Spinal Cord Stimulation — Non-invasive spinal cord stimulation will be applied. The resulting torque data will be collected, and ultrasound data will be obtained during stimulation.
Device: Ultrasound — Ultrasound data will be collected from the shin muscles during FES and tSCS.

SUMMARY:
Transcutaneous (non-invasive) spinal cord stimulation (tSCS) has been shown to facilitate volitional motor activity in patients with spinal cord injury. tSCS is known to activate the same neural structures as invasive SCS, meaning it may have the potential for functional restoration without an expensive surgical implant. Functional electrical stimulation (FES) is also used in therapy for patients with spinal cord injury to locally activate paralyzed or weakened muscles. There is evidence that combining FES and tSCS may elicit greater muscle activation than either modality alone.

The objective of this study is to quantify the torque at the ankle joint generated by tSCS, by FES, and by tSCS + FES. Additionally, ultrasound images will be collected during stimulation to provide a metric of muscle activity. The correlation between ultrasound and torque will be assessed to determine if ultrasound is a useful modality for quantifying tSCS-elicited muscle activity.

ELIGIBILITY:
Inclusion Criteria:

* Between 18 and 60 years of age
* Weight less than 220 lb
* Healthy and able to walk at preferred speed without an assistive device
* Able to tolerate functional electrical stimulation and tSCS.

Exclusion Criteria:

* Active infection
* history of cancer,
* broken skin, sores, or areas of acute eczema near the electrode sites
* metal implants, such as staples or pins, near the electrode sites
* any neurological disorders
* difficulty walking or an orthopedic condition that would impede walking normally without assistance
* absent sensation in the lower extremities or trunk (torso),
* allergies to adhesive skin tapes and/or ultrasound gels,
* heart conditions
* an implanted electronic device such as a pacemaker
* current pregnancy
* having no physiological response to FES and/or tSCS.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Ankle Joint Torque | Through study completion, estimated 12 months
  Ankle joint torque will be collected during stimulation with FES, with tSCS, and with FES + tSCS. We will compare the torque elicited by each simulation case.
Ultrasound-Derived Muscle Activation | Through study completion, estimated 12 months
  Ultrasound data will be collected from the shin muscles during FES, tSCS, and FES + tSCS. Muscle activation will be extracted from this data, and activation levels will be compared across stimulation cases.

CONTACTS AND LOCATIONS:
Locations (1):
- Engineering Building III, Raleigh, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared outside of this research group. However, selected data may be published in academic journals, conference papers, or other publications. This data will be de-identified, and will not include the full set of data.